CLINICAL TRIAL: NCT01512459
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-sequence Two-period, Single Dose Sprinkled on Apple Sauce, Crossover and Relative Bioavailability Study in Healthy Adult, Human Subjects Under Fed Conditions
Brief Title: Bioavailability Study of Venlafaxine MR Capsules 150 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 610/06
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Bioavailability; Venlafaxine; two way crossover
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venlafaxine MR Capsules 150 (Experimental): Venlafaxine MR Capsules 150 of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Venlafaxine
- Effexor XR 150 mg Capsules (Active Comparator): Effexor XR 150 mg Capsules of Wyeth Laboratories Philadelphia, PA, USA
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxine MR Capsules 150 mg
  Other Names: Effexor XR

SUMMARY:
The objective of this study was to compare the relative bioavailability of Venlafaxine MR Capsules 150 mg with Effexor XR Capsules 150 mg under Fed conditions in healthy adult human subjects.

DETAILED DESCRIPTION:
An open labeL balanced, randomized, two-treatment. two-period, two-sequence, single dose,crossover, evaluation of relative bioavailability of Venlafaxine 150 mg (as the HCl salt)MR capsules of Dr. Reddy's comparing with that of Effexor XR (containing Venlafaxine 150 mg (as the HCl salt)capsules of wyeth Laboratories, Philadelphia, PA, USA in healthy human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

* Subjects who will provide written informed consent.
* Subjects must be healthy human beings within 18-45 years of age (inclusive) weighing at least 50 kg.
* Having a Body mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2
* Subjects must be of normal health as determined by medical history and physical examination performed within 21days prior to the commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/investigator to be of no clinical significance.
* Have normal ECG, X-ray and vital signs.
* Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidence by written informed consent.

Exclusion Criteria:

* Subjects incapable of understanding the informed consent.
* Subjects who have:

  * Systolic blood pressure less than 90 mm of Hg and more than 140 .mm of Hg
  * Diastolic blood pressure less than 60 mm of Hg and more than 94 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the physician/investigator.
  * Pulse rate below 50/min and above 100/min.
* History of hypersensitivity or idiosyncratic reaction to Venlafaxine or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal .function.
* Consumption of grapefruit for the past ten days prior to the dosing day until the completion of the study.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and until the completion of the study.
* Subjects who have taken over the counter or prescribed medications for during the last 7 days from the date of study.
* Subjects who have taken enzyme modifying drugs or any systemic medication within the past 30 days prior to start of clinical study
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 330 mL in the past 90 days before the date of start of study.
* Subjects with positive screen for drugs of abuse and alcohol.
* Any subject in whom Venlafaxine is contraindicated for medical reasons.
* Any subject with recent history of surgery
* A history of difficulty in donating blood.
* A positive test result for HIV antibody and/or syphilis
* A recent history of alcoholism (< 2 years) or of moderate (180 ml/day) alcohol use, or consumption of alcohol within 48 hr prior to receiving Investigational Product.
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | predose, 1.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 9.00, 10.00, 12.00, 14.00, 24.00, 36.00, 48.00 and 72.00 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Mohanlal Siva Prasad Sayana, Dr., Principal Investigator — Bioserve Clinical Research (P) Ltd
Locations (1):
- Bioserve Clinical Research (P) Ltd, Bālānagar, Hyderabad, India